CLINICAL TRIAL: NCT00751556
Title: An Open Label, Randomized, Two-Way Crossover Trial to Determine the Pharmacokinetic Profile of an Extended Release Naproxen Sodium Tablet Relative to Aleve Tablets Following Single and Multiple Dose Administration in Healthy Adult Subjects
Brief Title: Single/Multiple Dose Bioavailability Trial
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 13106
Record Dates: First submitted 2008-09-11; First posted 2008-09-12 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Healthy
Keywords: Naproxen Sodium; Bioavailability
MeSH Terms: interventions — Naproxen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Naproxen Sodium 660mg
- Arm 2 (Active Comparator)
  Interventions: Drug: Commercial Aleve 220 mg

INTERVENTIONS:
Drug: Naproxen Sodium 660mg — Extended release Naproxen Sodium (660mg) administered once a day
  Arms: Arm 1
Drug: Commercial Aleve 220 mg — Immediate release commercial Aleve (220 mg) administered in a 2 (440 mg) plus one (220 mg) dosing schedule, 660 mg total
  Arms: Arm 2

SUMMARY:
To determine the pharmacokinetic profile of an extended release tablet of naproxen sodium 660 mg relative to the established commercial Aleve 220 mg tablet following single dose administration and at steady-state following multiple dose administration for 4 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, ambulatory, male and female volunteers between 18 - 55 years of age with BMI of approximately 18 to 30 kg/m2, and total body weight >50 kg (110Ibs)

Exclusion Criteria:

* History of hypersensitive to aspirin (ASA), naproxen sodium, or acetaminophen, and similar pharmacological agents or components of the products
* History of gastrointestinal bleeding or perforation related to previous Non-Steroidal Anti-Inflammatory Drug (NSAID) therapy Active, or history of current peptic ulcer/hemorrhage (two or more distinct episodes of proven ulceration or bleeding)
* Have taken ASA, ASA-containing products, acetaminophen (acetyl-para-amino-phenol or APAP) or any other NSAID (OTC or prescription) 7 days prior to dosing or during the treatment period, other than study treatment

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2008-02; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics parameters | Over 48 Hours

SECONDARY OUTCOMES:
Assess the safety and tolerability of the investigational product | Over 48 Hours

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Little Rock, Arkansas, United States